CLINICAL TRIAL: NCT07313280
Title: Psychological Profile Associated With the Complexity of Central Sensitization Syndromes, Comorbid With Trauma and Post-Traumatic Stress Disorder in Women: Testing the Effectiveness of a Person-Centered Psychological Intervention
Brief Title: Central Sensitization Syndromes and Post-Traumatic Stress in Women: Psychological Profile and Intervention
Acronym: SINSENTRA
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Collaborators: Ministerio de Ciencia, Innovación y Universidades, Spain (Unknown)
Responsible Party: Principal Investigator, Elena R. Serrano-Ibáñez, Principal Investigator, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PID2023-152784OA-I00
Record Dates: First submitted 2025-12-03; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Posttraumatic Stress Symptom; Central Sensitization; Chronic Pain Syndrome
Keywords: Central Sensitivity Syndromes; Post-traumatic stress; Chronic pain; Treatment
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: Study 2 will undertake an empirical investigation employing a manipulative strategy within an experimental design.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Profile 1_Reactive (Experimental): The arms will be developed based on the psychological profile identified in Study 1, given that a better understanding of CSS-PTSD comorbidity is necessary to design an effective intervention targeting the specific variables maintaining this condition.
  Interventions: Behavioral: CSS-PTSD psychological interventions
- Profile 2_Dysphoric (Experimental): The arms will be developed based on the psychological profile identified in Study 1, as a better understanding of CSS-PTSD comorbidity is necessary to design an effective intervention targeting the specific variables that maintain this condition.
  Interventions: Behavioral: CSS-PTSD psychological interventions
- Profile 3_Dissociative (Experimental): The arms will be developed based on the psychological profile identified in Study 1, given that a better understanding of CSS-PTSD comorbidity is necessary to design an effective intervention targeting the specific variables maintaining this condition.
  Interventions: Behavioral: CSS-PTSD psychological interventions
- Profile 4_Mixed (Experimental): The arms will be developed based on the psychological profile identified in Study 1, as a better understanding of CSS-PTSD comorbidity is necessary to design an effective intervention targeting the specific variables that maintain this condition.
  Interventions: Behavioral: CSS-PTSD psychological interventions

INTERVENTIONS:
Behavioral: CSS-PTSD psychological interventions — The interventions will be developed based on the techniques previously developed within cognitive behavioural approaches, which have demonstrated efficacy in treating both conditions.

SUMMARY:
Central Sensitivity Syndromes (CSSs) are a group of conditions that are highly prevalent, particularly among women, and often occur alongside post-traumatic stress disorder (PTSD).

This research project has two aims: Study 1) to investigate the psychological profiles of women with CSS-PTSD comorbidity; and Study 2) to design and evaluate the effectiveness of distinct interventions for each profile identified in Study 1.

DETAILED DESCRIPTION:
Central Sensitivity Syndromes (CSSs) are a group of conditions, including fibromyalgia and chronic pelvic pain, associated with symptoms such as perceived pain intensity, depression, anxiety, stress, sleep disturbances, and disability. These syndromes are highly prevalent, particularly among women, and often occur alongside post-traumatic stress disorder (PTSD). This condition stems from a variety of traumatic experiences and manifests as a range of symptoms in individuals with different psychological profiles. However, not all individuals who experience trauma develop PTSD or CSSs, nor do all individuals with CSSs have PTSD or exhibit the same symptom patterns. Transdiagnostic psychological variables may contribute to the development and maintenance of both conditions. Commonly observed factors in both CSSs and PTSD include emotional dysregulation, anxiety sensitivity, experiential avoidance, distress intolerance, and dissociation. These transdiagnostic vulnerability variables could be associated with each profile. Identifying these profiles may enable targeted interventions that address the underlying vulnerabilities driving CSS-PTSD comorbidity. By aligning treatment to individual vulnerability patterns, this approach aims to improve outcomes for women affected by CSS-PTSD.

Four PTSD profiles will be identified:

* Reactive (with prominent intrusions, avoidance, and hyperarousal).
* Dysphoric (with anhedonia and negative affect).
* Dissociative (with high negative and positive dissociative symptoms).
* Mixed (with high levels of all PTSD symptoms). However, no studies have analysed how these transdiagnostic vulnerability variables (emotion dysregulation, anxiety sensitivity, experiential avoidance, distress intolerance, and dissociation) are grouped and shape the different PTSD symptom profiles in populations with either PTSD or comorbid CSS. Therefore, the analysis of the association between PTSD profiles and transdiagnostic variables is exploratory.

The treatments will be developed based on the variables associated with each profile identified in Study 1.

ELIGIBILITY:
Inclusion Criteria:

1. being a biological woman.
2. having a medical diagnosis of CSS.
3. scoring >36 on the Posttraumatic Stress Disorder Checklist for DSM-5, which indicates PTSD in people with chronic pain.
4. having the ability to understand and sign the informed consent form.

Exclusion Criteria:

1. having a diagnosis of serious mental illness or neurodegenerative disease.
2. not being fluent in spoken and written Spanish.
3. undergoing treatment for an oncological, degenerative, or terminal disease.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-10-02 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in anxiety sensitivity | Pre-treatment (T1), Post-treatment (T2; 24 weeks after T1), 3-months follow-up (T3), 6-months follow-up (T4).
  The Spanish version of the Anxiety Sensitivity Index (ASI-3). It is a 16-item questionnaire; items are rated from 0 ("Not at all or almost nothing) to 4 ("Very much"), with higher total scores indicating greater anxiety sensitivity.
Change in emotion dysregulation | Pre-treatment (T1), Post-treatment (T2; 24 weeks after T1), 3-months follow-up (T3), 6-months follow-up (T4).
  The Spanish brief version of the Difficulties in Emotion Regulation Scale (DERS-S SF). It comprises 18 items with a 5-point Likert scale, from 1("Almost never) to 5 "Almost always") divide into 5 subscales: nonacceptance of emotional responses, difficulty engaging in goal-directed behaviour, impulse control difficulties, limited access to emotion regulation strategies, and lack of emotional clarity. Higher total scores indicate greater difficulties in emotion regulation.
Change in experiential avoidance | Pre-treatment (T1), Post-treatment (T2; 24 weeks after T1), 3-months follow-up (T3), 6-months follow-up (T4).
  The Spanish version of the Acceptance and Action Questionnaire II (AAQ II). It is a brief 7-item instrument; items are a 7-point Likert-type scale, ranging from 1 ("Never") to 7 ("Always"). Higher total scores indicate greater experiential avoidance.
Change in distress intolerance | Pre-treatment (T1), Post-treatment (T2; 24 weeks after T1), 3-months follow-up (T3), 6-months follow-up (T4).
  The Spanish version of the Distress Tolerance Scale (DTS). It is a 15-item questionnaire; items are rated from 1 ("Strongly agree") to 5 ("Strongly disagree"), with higher total scores indicating greater distress tolerance.
Change in dissociative symptoms | Pre-treatment (T1), Post-treatment (T2; 24 weeks after T1), 3-months follow-up (T3), 6-months follow-up (T4).
  The Spanish version of the abbreviated scale of the Dissociative Experiences Scale-Modified (DES-M). It consists of 18 questions, rated on a 5-point Likert-type scale (ranging from 1 = "Never" to 5 = "Always"), with higher total scores indicating greater dissociative symptoms.
Change in daily symptom monitoring | Treatment (periprocedural), 1-months follow-up.
  Participants will complete an electronic diary from the time of the initial assessment until 30 days post-intervention.
  Electronic diary developed and validated by Åkerblom et al., 2022.

SECONDARY OUTCOMES:
Change in Central Sensitization Indexes | Pre-treatment (T1), Post-treatment (T2; 24 weeks after T1), 3-months follow-up (T3), 6-months follow-up (T4).
  1. Spanish Central Sensitization Inventory (CSI). It is a 25-item questionnaire that comprises a 5-point Likert scale, ranging from 0 ('Never') to 4 ('Always'). Higher total scores indicate greater central sensitization symptoms.
  2. Quantitative sensory testing (QST). Tests that allow the nociceptive system to be comprehensively evaluated and obtain objective information on how pain is perceived.
Change in posttraumatic stress symptoms | Pre-treatment (T1), Post-treatment (T2; 24 weeks after T1), 3-months follow-up (T3), 6-months follow-up (T4).
  The Spanish version of the Posttraumatic Stress Disorder Checklist-5 (PCLC-5). A 20-item self-report, with a Likert-type scale ranging from 1 ("Not at all") to 5 ("Very much"). Higher total scores indicate greater posttraumatic stress symptoms.
Change in stress symptoms | Pre-treatment (T1), Post-treatment (T2; 24 weeks after T1), 3-months follow-up (T3), 6-months follow-up (T4).
  Stress subscale of the Depression Anxiety Stress Scale (DASS-21). It is a 7-item subscale; items are rated from 0 ("Never") to 3 ("Almost always"), with higher total scores indicating greater stress symptoms.
Change in anxiety and depressive symptoms | Pre-treatment (T1), Post-treatment (T2; 24 weeks after T1), 3-months follow-up (T3), 6-months follow-up (T4).
  The Spanish version of the Hospital Anxiety and Depression Scale (HADS). It has two subscales (Anxiety and Depression) with 7 questions each, scored 0-3, totaling 0-21 per subscale, where higher scores indicate greater severity
Change in sleep disturbance | Pre-treatment (T1), Post-treatment (T2; 24 weeks after T1), 3-months follow-up (T3), 6-months follow-up (T4).
  The Spanish version of PROMIS 8b-item Sleep Disturbance Scale. It uses 8 questions to assess difficulty falling/staying asleep, restlessness, and satisfaction, scored on a 5-point Likert scale (from 1 = "Never" to 5 = "Always"), with higher scores indicating worse sleep quality.
Change in pain interference | Pre-treatment (T1), Post-treatment (T2; 24 weeks after T1), 3-months follow-up (T3), 6-months follow-up (T4).
  The Short Form of the Brief Pain Inventory (BPI-SF). A 9-item self-report questionnaire assessing pain severity (worst, least, average, current) and its interference with daily life (activity, mood, sleep, work, etc.); items are rated from 0 ("no pain"/"not interferes") to 4 ("worst pain imaginable" /"completely interferes"), with higher total scores indicating greater pain interference.

OTHER OUTCOMES:
Adverse Events (side effects) | Treatment (periprocedural) and 3-months follow-up, 6-months follow-up.
  Adverse Events are not expected given the content of the treatment and its non-invasive nature, however, they will be assessed, recorded and controlled for in the analyses.
Change in medical data | Pre-treatment (T1), Post-treatment (T2; 24 weeks after T1), 3-months follow-up (T3), 6-months follow-up (T4).
  Medication intake (analgesics and psychotropic drugs), dose, and healthcare utilization.

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Hospital Universitario Regional de Málaga_Hospital Civil, Málaga, Málaga
  - Hospital Universitario Virgen de la Victoria, Málaga, Málaga
  - Área de Gestión Sanitaria Este de Málaga-Axarquía, Málaga, Torre Del Mar

IPD SHARING:
Plan to Share IPD: No